CLINICAL TRIAL: NCT00121004
Title: A Study to Tailor Advance Directives
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13787A
Record Dates: First submitted 2005-07-11; First posted 2005-07-19 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Dementia; Persistent Vegetative State; Terminally Ill
Keywords: Advance Directive; Living Will; Terminal Illness
MeSH Terms: conditions — Dementia; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Advance Directive Selection

SUMMARY:
In this study, hospitalized patients will first be surveyed regarding their interest in a traditional advanced directive (AD) and then in a modified AD.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether patients will execute an advance directive which offers a limited trial of life-sustaining therapy in non-terminal illness, declines life-sustaining therapy or artificial nutrition in advanced dementia, or declines life-sustaining therapy in general. Advance directives (ADs) as currently drafted have been questioned since they have not had much effect on end-of-life care. However, the reason for the lack of success may be simply that they rarely apply. Traditional ADs, which are limited to terminal illness or persistent vegetative states, are difficult to apply to the more common cases of critical illness in the setting of potentially reversible disease and advanced dementia, which are often not recognized as terminal. In addition, terminal ADs are drafted too narrowly for patients who do not wish for life-sustaining therapy regardless of condition.

Patients may execute either AD at the conclusion of the survey. This research has the potential to demonstrate widely reproducible methods on which more precise advance planning can be based and thereby improve end-of-life care.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients admitted to the general medical service at the University of Chicago
* Previously enrolled in a study of hospitalized general medicine patients at the University of Chicago

Exclusion Criteria:

* Patients who score less than 17 out of 30 on the Folstein Mini-Mental Status Examination or who have a proxy decision-maker
* Patients who are medically unstable based on two or more abnormal vital signs
* Patients who face a possible new diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients admitted to the general medical service at the University of Chicago
Sampling Method: Non-Probability Sample
Enrollment: 100
Dates: Start 2005-07; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elmer Abbo, M.D., Ph.D., Principal Investigator — University of Chicago; David Meltzer, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] A controlled trial to improve care for seriously ill hospitalized patients. The study to understand prognoses and preferences for outcomes and risks of treatments (SUPPORT). The SUPPORT Principal Investigators. JAMA. 1995 Nov 22-29;274(20):1591-8. PMID 7474243
- [Background] Teno JM, Licks S, Lynn J, Wenger N, Connors AF Jr, Phillips RS, O'Connor MA, Murphy DP, Fulkerson WJ, Desbiens N, Knaus WA. Do advance directives provide instructions that direct care? SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatment. J Am Geriatr Soc. 1997 Apr;45(4):508-12. doi: 10.1111/j.1532-5415.1997.tb05179.x. PMID 9100722
- [Background] Teno JM, Lynn J, Phillips RS, Murphy D, Youngner SJ, Bellamy P, Connors AF Jr, Desbiens NA, Fulkerson W, Knaus WA. Do formal advance directives affect resuscitation decisions and the use of resources for seriously ill patients? SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. J Clin Ethics. 1994 Spring;5(1):23-30. No abstract available. PMID 8003719
- [Background] Danis M, Southerland LI, Garrett JM, Smith JL, Hielema F, Pickard CG, Egner DM, Patrick DL. A prospective study of advance directives for life-sustaining care. N Engl J Med. 1991 Mar 28;324(13):882-8. doi: 10.1056/NEJM199103283241304. PMID 2000110
- [Background] Schneiderman LJ, Kronick R, Kaplan RM, Anderson JP, Langer RD. Effects of offering advance directives on medical treatments and costs. Ann Intern Med. 1992 Oct 1;117(7):599-606. doi: 10.7326/0003-4819-117-7-599. PMID 1524334
- [Background] Ditto PH, Danks JH, Smucker WD, Bookwala J, Coppola KM, Dresser R, Fagerlin A, Gready RM, Houts RM, Lockhart LK, Zyzanski S. Advance directives as acts of communication: a randomized controlled trial. Arch Intern Med. 2001 Feb 12;161(3):421-30. doi: 10.1001/archinte.161.3.421. PMID 11176768
- [Background] Fagerlin A, Schneider CE. Enough. The failure of the living will. Hastings Cent Rep. 2004 Mar-Apr;34(2):30-42. PMID 15156835
- [Background] Miles SH, Koepp R, Weber EP. Advance end-of-life treatment planning. A research review. Arch Intern Med. 1996 May 27;156(10):1062-8. PMID 8638992
- [Background] Teno JM. Advance directives: time to move on. Ann Intern Med. 2004 Jul 20;141(2):159-60. doi: 10.7326/0003-4819-141-2-200407200-00017. No abstract available. PMID 15262674
- [Background] Lunney JR, Lynn J, Hogan C. Profiles of older medicare decedents. J Am Geriatr Soc. 2002 Jun;50(6):1108-12. doi: 10.1046/j.1532-5415.2002.50268.x. PMID 12110073
- [Background] Fried TR, Bradley EH, Towle VR, Allore H. Understanding the treatment preferences of seriously ill patients. N Engl J Med. 2002 Apr 4;346(14):1061-6. doi: 10.1056/NEJMsa012528. PMID 11932474
- [Background] Danis M, Patrick DL, Southerland LI, Green ML. Patients' and families' preferences for medical intensive care. JAMA. 1988 Aug 12;260(6):797-802. PMID 3392810
- [Background] Starr TJ, Pearlman RA, Uhlmann RF. Quality of life and resuscitation decisions in elderly patients. J Gen Intern Med. 1986 Nov-Dec;1(6):373-9. doi: 10.1007/BF02596420. PMID 3794836
- [Background] Silverstein MD, Stocking CB, Antel JP, Beckwith J, Roos RP, Siegler M. Amyotrophic lateral sclerosis and life-sustaining therapy: patients' desires for information, participation in decision making, and life-sustaining therapy. Mayo Clin Proc. 1991 Sep;66(9):906-13. doi: 10.1016/s0025-6196(12)61577-8. PMID 1921500
- [Background] Murphy DJ, Santilli S. Elderly patients' preferences for long-term life support. Arch Fam Med. 1998 Sep-Oct;7(5):484-8. doi: 10.1001/archfami.7.5.484. PMID 9755744
- [Background] Blackhall LJ, Frank G, Murphy ST, Michel V, Palmer JM, Azen SP. Ethnicity and attitudes towards life sustaining technology. Soc Sci Med. 1999 Jun;48(12):1779-89. doi: 10.1016/s0277-9536(99)00077-5. PMID 10405016
- [Background] Gjerdingen DK, Neff JA, Wang M, Chaloner K. Older persons' opinions about life-sustaining procedures in the face of dementia. Arch Fam Med. 1999 Sep-Oct;8(5):421-5. doi: 10.1001/archfami.8.5.421. PMID 10500515
- [Background] Robertson GS. Resuscitation and senility: a study of patients' opinions. J Med Ethics. 1993 Jun;19(2):104-7. doi: 10.1136/jme.19.2.104. PMID 8080470
- [Background] Emanuel LL, Barry MJ, Stoeckle JD, Ettelson LM, Emanuel EJ. Advance directives for medical care--a case for greater use. N Engl J Med. 1991 Mar 28;324(13):889-95. doi: 10.1056/NEJM199103283241305. PMID 2000111
- [Background] Lo B, McLeod GA, Saika G. Patient attitudes to discussing life-sustaining treatment. Arch Intern Med. 1986 Aug;146(8):1613-5. No abstract available. PMID 3729645
- [Background] Singer PA, Thiel EC, Salit I, Flanagan W, Naylor CD. The HIV-specific advance directive. J Gen Intern Med. 1997 Dec;12(12):729-35. doi: 10.1046/j.1525-1497.1997.07157.x. PMID 9436891
- [Background] Griffith CH 3rd, Wilson JF, Emmett KR, Ramsbottom-Lucier M, Rich EC. Knowledge and experience with Alzheimer's disease. Relationship to resuscitation preference. Arch Fam Med. 1995 Sep;4(9):780-4. doi: 10.1001/archfami.4.9.780. PMID 7647944
- [Background] Everhart MA, Pearlman RA. Stability of patient preferences regarding life-sustaining treatments. Chest. 1990 Jan;97(1):159-64. doi: 10.1378/chest.97.1.159. PMID 2104791
- [Background] Berger JT, Majerovitz D. Stability of preferences for treatment among nursing home residents. Gerontologist. 1998 Apr;38(2):217-23. doi: 10.1093/geront/38.2.217. PMID 9573666
- [Background] Mitchell SL, Kiely DK, Hamel MB. Dying with advanced dementia in the nursing home. Arch Intern Med. 2004 Feb 9;164(3):321-6. doi: 10.1001/archinte.164.3.321. PMID 14769629